CLINICAL TRIAL: NCT02327065
Title: Prospective Multi-center, Single Blinded, Randomized, Controlled Trial of EUS-FNB（Endoscopic Ultrasonography-Fine Needle Biopsy ） and EUS-FNA（Endoscopic Ultrasonography-Fine Needle Aspiration ） on Solid Occupying Lesion
Brief Title: Prospective Multi-center, Single Blinded, Randomized, Controlled Trial of EUS-FNB and EUS-FNA on Solid Occupying Lesion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Bin Cheng, professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2014tj1212
Record Dates: First submitted 2014-12-11; First posted 2014-12-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Pancreas Neoplasms; Lymphatic Metastasis; Neoplasm Metastases; Unknown Primary Neoplasm Metastasis
Keywords: EUS; FNA; FNB
MeSH Terms: conditions — Pancreatic Neoplasms; Lymphatic Metastasis; Neoplasm Metastasis; Neoplasms, Unknown Primary | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EUS-FNA Group (Active Comparator): FNA,Fine needle aspiration
  Interventions: Device: EUS-FNA (EchoTip Ultra)
- EUS-FNB Group (Active Comparator): FNB,Fine needle biopsy
  Interventions: Device: EUS-FNB (EchoTip ProCore)

INTERVENTIONS:
Device: EUS-FNA (EchoTip Ultra) — FNA,Fine needle aspiration
  Other Names: EchoTip Ultra needle
  Arms: EUS-FNA Group
Device: EUS-FNB (EchoTip ProCore) — FNB,Fine needle biopsy
  Other Names: EchoTip ProCore needle
  Arms: EUS-FNB Group

SUMMARY:
The purpose of this study is to compare the diagnosis accuracy of FNA and FNB biopsy on pancreatic, retroperitoneal, mediastinum and pelvic cavity solid occupying lesions.

DETAILED DESCRIPTION:
The study subjects are divided into two groups: the EUS-FNA(22G EchoTip Ultra needles) Group and EUS-FNB group(22G EchoTip ProCore needles).Take the malignant occupying lesion diagnosis accuracy as the research major indicator to compare the EUS-FNB group and EUS-FNA group as optimal efficiency test. Take the class I error a=0.05, class II error β=0.15, power=0.85. Suppose the malignancy diagnosis accuracy is 80%, while that of FNB is 93%. The two trial groups be randomly allocated in 1:1, suppose the malignancy cases take 70% of the whole case, and considering the shedding factors , extra 20% cases should be included. So the estimated cases numbers is 204 cases for EUS-FNB group and 204 cases for EUS-FNA group, totally 408 cases in this trial.

Done by professional statistical people with randomized block grouping method and SAS 9.2 statistical software to generate randomized serial number（001-408）for the two groups in 1:1 manner. The serial numbers are the randomized grouping numbers for the trial patients, block capacity is 8, totally 51 randomized block. The randomized grouping will be generated in duplicate copies and sealed. One copy send to trial centers for patient allocating, and the another copy be saved by the trial applicant unit. Every trail centers will be responsible for the screening of qualified patients, rank them in visit time to get the randomized grouping number so as to determine them goes to the EUS-FNA or EUS-FNB.The research people and patients in all trial centers should not know the the randomized grouping number and relevant groups. The group name will be sealed under scratch card. Every trial patients will get a unique randomized number, and it will not change through out the whole trial.

Use the inclusion and exclusion criteria to observe the patients and do relative inspections, and confirm if the patients qualified or not to the trial. Record the result of last time test before the treatment. Although it is better to get the informed consent before doing all kinds of observation and tests, if for some reason, the medical imaging examination has completed, as long as the imaging examination was done within 3 weeks before the needle biopsy, it can still be collect as baseline data (imaging examination can be done at other hospitals, but the trial center should issue a new evaluation report 1 week before the patient join the trial group); other lab test items done at 2 weeks before the needle biopsy can still be collect as baseline data for pre-research use, but these tests should be done at the trail center hospital so as to guarantee the data trace ability.

The investigators will do the needle passes for 4 times for all of them:the 1-2 needle passes with Slow-Pull and the 3-4 needle passes with Vacuum suction.If no core tissues obtained or the operator/onsite pathologist determine insufficient specimen after the operations above, then remedy procedures will be done, the operator use proper puncture method to continue the remedy biopsy.After the first round of needle biopsy, if the trial patient cannot be diagnosed, by getting the agreement of the patient, the patient will be cross-over to another trial group and do needle biopsy again on the same lesion 1 week later with the method mentioned above.Without knowing the needle biopsy type, the cytologist and pathologist evaluate the specimen quality and make diagnosis. Every specimen will be independently evaluated and diagnosed by 2 experts. If the 2 experts have different judgments, then these two experts discuss together and make the final diagnose discussion. If the same sample has 2 or more cytology smear slides, than take the highest score slide as the result.Follow up (outpatient follow up or telephone follow up) the patients at 1 week, 12 weeks and 36 weeks after the needle biopsy and collect the patients clinical data and confirm their final diagnosis.

During the trial, if severe adverse event occurs, the trialed center must take immediate actions necessary to guarantee the trialed patients' safety. Once severe adverse event occurs, the researchers should inform the trial applicant and the trail center's ethics committee within 24 hours after the researchers gets to know the adverse event. And the researchers should also fax the report to State Food and Drug Administration of China and the local provincial food and drug administration. After receiving the report, the applicant should inform other clinical trial centers within 24 hours. All the severe adverse events should be filed at group leader medical center and other trial centers.

CRF(Case Report Form ) will be filled by the researchers, every involved patient must have the CRF(Case Report Form ) filled. This will be audited by clinical monitor and handed over to data administrator to input and manage data, the first copy will be kept by the applicant, the second copy will go to the trial center, and the third copy will be kept by the trail researchers.The data input and management will be taken care by specially assigned person. In order to guarantee the data accuracy, data input will be done twice by two independent data administrators, by computerized and manual verifying, hand over the data to statistical experts to do blind check and statistic analyzing.For the questions and doubts within the case report form, the data administrator make DRQ and via the clinical monitor asking the researchers. The researchers will answer and feed back as soon as possible. According to the researchers answer, data administrator will do the data modifying, confirming or inputting, and when necessary send out DRQ again.After blind audition and confirming that the established data base is correct, major researchers, applicant and the statistic analyzing people lock the data. The locked data will not be changed, and the data base will be handed over to statistical analyzer to do the statistic analyze according to the statistic analyzing plan. Problems found after data locking can be modified during the statistic analyzing procedure.This will be done by specialized statistic analyzing people according to the predetermined statistic analyzing plan. The statistic analyze will be carried out according to intention principle confirmed full analysis set and per-protocol set principle. After completing the statistic analyzing, the statistic analyzer issue the statistic analysis report and send this to major researchers to write the study report.

Statistic analyzing plan:⑴ General principle:① all the statistic tests are use the two-tailed-test method, P<0.05 will be thought as the tested difference is statistical significance. ② the quantitative indicator description will calculate the Mean and Standard deviation. The classification indicator description will describe the cases and percentage of all types of cases. ⑵ Statistic analyzing method:① for the measurement data, compare it with the baseline value at selection period, use paired t-test or symbol rank sum test to compare with the before-after-difference within the group.② for the counting data, use x2 test to compare the groups. ⑶ Shedding analysis:Comparison of groups'total shedding rates and the shedding rates caused by adverse events will use x2 test or Fisher's exact test method. ⑷ The baseline value's equilibrium analysis: Use group t test or x2 test to compare the demography info and vital signs, disease history, and basic treatment and other indicators of baseline value, so as to measure the balance of the groups. The baseline evaluation will be done on FAS（full analysis set) and PPs(per-protocol set). ⑸ Effectiveness analysis:The major indicator of effectiveness analysis is the diagnostic accuracy on malignant disease, and the indicators of second effectiveness include the percentage of Grade A specimen and complications rate etc. while the two groups rate and the Youden index comparison will use approximate normal Z test or use central effect x2 test.(6) Safety analysis:Use x2 test or Fisher's exact test to compare the adverse event/adverse reaction (include biopsy complications) rates between the groups. And use table to describe the adverse events during this trial project; the lab test results before and after the trial, the normal/abnormal changing condition and the relationship with this trial research when abnormal changes happened.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred for EUS tissue sampling who provide informed consent

Exclusion Criteria:

* Coagulopathy which is not corrected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-08 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Yield on malignancy | 18 months
  The investigators' primary outcome measure is to compare the the diagnostic yield (%) on malignancy of EUS-FNA to EUS-FNB

SECONDARY OUTCOMES:
Blood contamination and cellularity in specimens obtained by EUS-FNA and EUS-FNB with Slow-pull or suction | 18 months
  The amount of blood contamination and cellularity at each sample according to EUS-FNA and EUS-FNB with slow-pull or suction will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Bin Cheng, Doctor, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Result] DeWitt J, Jowell P, Leblanc J, McHenry L, McGreevy K, Cramer H, Volmar K, Sherman S, Gress F. EUS-guided FNA of pancreatic metastases: a multicenter experience. Gastrointest Endosc. 2005 May;61(6):689-96. doi: 10.1016/s0016-5107(05)00287-7. PMID 15855973
- [Result] Puli SR, Batapati Krishna Reddy J, Bechtold ML, Ibdah JA, Antillon D, Singh S, Olyaee M, Antillon MR. Endoscopic ultrasound: it's accuracy in evaluating mediastinal lymphadenopathy? A meta-analysis and systematic review. World J Gastroenterol. 2008 May 21;14(19):3028-37. doi: 10.3748/wjg.14.3028. PMID 18494054
- [Result] Puri R, Vilmann P, Sud R, Kumar M, Taneja S, Verma K, Kaushik N. Endoscopic ultrasound-guided fine-needle aspiration cytology in the evaluation of suspected tuberculosis in patients with isolated mediastinal lymphadenopathy. Endoscopy. 2010 Jun;42(6):462-7. doi: 10.1055/s-0029-1244133. Epub 2010 Apr 29. PMID 20432206
- [Result] Wiersema MJ, Vilmann P, Giovannini M, Chang KJ, Wiersema LM. Endosonography-guided fine-needle aspiration biopsy: diagnostic accuracy and complication assessment. Gastroenterology. 1997 Apr;112(4):1087-95. doi: 10.1016/s0016-5085(97)70164-1. PMID 9097990
- [Result] Gress FG, Hawes RH, Savides TJ, Ikenberry SO, Lehman GA. Endoscopic ultrasound-guided fine-needle aspiration biopsy using linear array and radial scanning endosonography. Gastrointest Endosc. 1997 Mar;45(3):243-50. doi: 10.1016/s0016-5107(97)70266-9. PMID 9087830
- [Result] Affolter KE, Schmidt RL, Matynia AP, Adler DG, Factor RE. Needle size has only a limited effect on outcomes in EUS-guided fine needle aspiration: a systematic review and meta-analysis. Dig Dis Sci. 2013 Apr;58(4):1026-34. doi: 10.1007/s10620-012-2439-2. Epub 2012 Oct 21. PMID 23086117
- [Result] Iglesias-Garcia J, Poley JW, Larghi A, Giovannini M, Petrone MC, Abdulkader I, Monges G, Costamagna G, Arcidiacono P, Biermann K, Rindi G, Bories E, Dogloni C, Bruno M, Dominguez-Munoz JE. Feasibility and yield of a new EUS histology needle: results from a multicenter, pooled, cohort study. Gastrointest Endosc. 2011 Jun;73(6):1189-96. doi: 10.1016/j.gie.2011.01.053. Epub 2011 Mar 21. PMID 21420083
- [Result] Lee JK, Choi JH, Lee KH, Kim KM, Shin JU, Lee JK, Lee KT, Jang KT. A prospective, comparative trial to optimize sampling techniques in EUS-guided FNA of solid pancreatic masses. Gastrointest Endosc. 2013 May;77(5):745-51. doi: 10.1016/j.gie.2012.12.009. Epub 2013 Feb 21. PMID 23433878
- [Result] Layfield LJ, Schmidt RL, Hirschowitz SL, Olson MT, Ali SZ, Dodd LL. Significance of the diagnostic categories "atypical" and "suspicious for malignancy" in the cytologic diagnosis of solid pancreatic masses. Diagn Cytopathol. 2014 Apr;42(4):292-6. doi: 10.1002/dc.23078. Epub 2014 Feb 28. PMID 24578254
- [Derived] Cheng B, Zhang Y, Chen Q, Sun B, Deng Z, Shan H, Dou L, Wang J, Li Y, Yang X, Jiang T, Xu G, Wang G. Analysis of Fine-Needle Biopsy vs Fine-Needle Aspiration in Diagnosis of Pancreatic and Abdominal Masses: A Prospective, Multicenter, Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2018 Aug;16(8):1314-1321. doi: 10.1016/j.cgh.2017.07.010. Epub 2017 Jul 19. PMID 28733257
- [Derived] Wang J, Wu X, Yin P, Guo Q, Hou W, Li Y, Wang Y, Cheng B. Comparing endoscopic ultrasound (EUS)-guided fine needle aspiration (FNA) versus fine needle biopsy (FNB) in the diagnosis of solid lesions: study protocol for a randomized controlled trial. Trials. 2016 Apr 12;17:198. doi: 10.1186/s13063-016-1316-2. PMID 27071386